CLINICAL TRIAL: NCT04887103
Title: The Effect of Hot Water Application in Pregnant Women With Restless Legs Syndrome: A Randomised Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ozlem Kaplan, Reserch Asistant, TC Erciyes University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Kaplan O-Erciyes University
Record Dates: First submitted 2021-05-12; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Restless Legs Syndrome; Pregnancy Related
Keywords: Restless legs syndrome; pregnancy; hot water application; nursing
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Intervention Model Description: pretest-posttest randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hot water application (Experimental): Pregnant women will apply hot water to their legs before going to sleep for a week.
  Interventions: Other: Hot water application
- Control group (No Intervention): There will be no intervention other than routine follow-up and maintenance.

INTERVENTIONS:
Other: Hot water application — Pregnant women will apply hot water to their legs before going to sleep for a week.
  Arms: hot water application

SUMMARY:
Backgraund and Purpose: The prevalance of restless legs syndrome (RLS) in pregnants varies between 15.4-26.0 percent. As well as pharmacological methods, there are studies reporting that non-pharmacological methods reduce RLS symptoms but the number of studies conducted with pregnants is limited. This study was conducted to determine the effect of hot water application to the legs of pregnants with RLS on their complaints.

Materials and methods: The study is a pretest-posttest randomised controlled. Among the pregnants whose IRLS score was more than 11, 13 people to the intervention group and 16 people to the control group were randomised. The data were collected using Personal Information Form, International RLS Study Group Diagnostic Criteria, and the International RLS Rating Scale (IRLS). Hot water application was made of intervention group. The application was made for 20 minutes before bedtime for seven days. No application was made in the control group other than routine care and follow-up. Chi-square test, descriptive statistics and dependent/independent samples t tests were used to assess the data. The value of p<0.05 was accepted as significant.

ELIGIBILITY:
Inclusion Criteria:

* in the gestation age of 28-32 weeks,
* literate,
* according to RLS Diagnostic Criteria and had 11 and higher severity according to International RLS Rating Scale (IRLS)

Exclusion Criteria:

* risky pregnancies,
* communication problems,
* any chronic and psychiatric disease
* were using antipsychotic, antidepressant, antihistaminic, and antiemetic drugs,
* had history of deep vein thrombosis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 29 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
RLS Severity Rating Scale | change from baseline score at the end of one week
  The RLS Severity Rating Scale was developed in 2003 by the International Restless Legs Syndrome Study Group. The scale was applied in the selection of patients and in the weekly evaluation of RLS severity. The scale comprised ten questions; each question was scored between 0 and 4. Questions 1, 2, 4, 6, 7, and 8 were related to RLS symptoms, questions 5, 9, and 10 were related to the effect of the disease on the mental state and daily social activities of patients with RLS, and question 3 was about the diagnostic criteria of RLS. The overall score indicated the RLS severity. A minimum score of 0 and a maximum score of 40 could be obtained. A score between 1 and 10 corresponded to "mild," 11-20 "moderate," 21-30 "severe," and 31-40 "very severe" RLS.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is thought to be shared after publication as an article.